CLINICAL TRIAL: NCT02673918
Title: The Breast Cancer Online Rehabilitation Program: A Feasibility Study of Individually Tailored Online Rehabilitation After Breast Cancer Surgery The Copenhagen BRECOR Program
Brief Title: The Breast Cancer Online Rehabilitation Program
Acronym: BRECOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Kristin Campbell, Associate Professor, University of British Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCCH-UBC 01
Record Dates: First submitted 2016-01-12; First posted 2016-02-04 (Estimated); Results first posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-11

CONDITIONS: Breast Cancer
Keywords: Rehabilitation; Home-Based Intervention
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This study was conducted in two parts and thereby had two groups of participants. Part 1 participants were newly operated for breast cancer. Part 2 participants had completed surgery and radiation therapy for breast cancer. Both groups received the same intervention, namely a home-based rehabilitation program.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1: Rehabilitation after surgery for breast cancer (Experimental): Home-based upper-body rehabilitation with online support
  Interventions: Other: Home-based upper-body rehabilitation with online support
- Part 2: Rehabilitation after radiation for breast cancer (Experimental): Home-based upper-body rehabilitation with online support
  Interventions: Other: Home-based upper-body rehabilitation with online support

INTERVENTIONS:
Other: Home-based upper-body rehabilitation with online support — Participants will be given written educational material, in which the physiotherapist marks the exercises specifically recommended for the individual patient. In addition, participants will get a personal password giving access to the BRECOR website for 12 weeks. The website contains professionally filmed videos of upper-body rehabilitation exercises (joint mobility and muscle strength) and instructions in scar tissue massage and manual lymph drainage. Furthermore, mindfulness sessions and additional information about prevention and early detection of late effects after breast cancer treatment are available on the website.
  On average, participants will complete three rehabilitation exercises 5-7 times weekly with an anticipated duration of approximately 20 minutes.

SUMMARY:
The investigators have developed an online rehabilitation platform to guide women in their home-based upper-body exercises after breast cancer surgery. The platform includes rehabilitation videos that will guide the women in performing home-based early post-surgery upper-body rehabilitation tailored for each individual.

The primary objective is to assess the feasibility and acceptability of a home-based rehabilitation program supported by a supplemental online platform for women after breast cancer surgery before conducting a larger pragmatic trial in the future. The feasibility of the platform will be tested in 11 municipalities in Denmark.

DETAILED DESCRIPTION:
More and more women are being diagnosed with breast cancer worldwide. While a vast majority will survive their disease, adverse treatment effects are common, and may persist beyond the treatment period and contribute to the burden of cancer. After surviving breast cancer, women often struggle with upper-body side effects from the cancer treatment such as tight scar tissue, arm swelling, decreased shoulder function. This limits the woman's physical well-being, affects her ability to take care of her family, return to work, and ultimately impacts her quality of life. Specific upper-body rehabilitation exercises and participation in general exercise have been shown to prevent, attenuate or rehabilitate many of the physical and psychosocial side effects of breast cancer treatment.

New ways of delivering rehabilitation are needed to ensure continued capacity to undertake the growing demand for cancer rehabilitation. There is currently great diversity in the quality and access to cancer rehabilitation. Equal access to evidence-based, homogeneous, and high-quality rehabilitation is needed independent of geographical area of residence and setting of rehabilitation (municipality or hospital).

Online rehabilitation integrated in the current survivorship rehabilitation programs offers the opportunity to deliver this homogeneous intervention across the country. At this time, little effort has been made to develop online rehabilitation platforms for breast cancer survivors, thus no evidence to support the expected benefits of online rehabilitation is available.

Study objective:

The study aims to test if the platform is feasible and acceptable for women who have received treatment for breast cancer. The hypothesis is that the support of filmed accessible upper-body rehabilitation exercises through a website will promote improved adherence and motivation to do the home-based exercises illustrated by ≥75% of participants will perform the home-based program 5-7 times weekly and ≥ 75% of participants report to be somewhat or very satisfied with the intervention.

Study design:

This study will test the feasibility of the intervention among two groups of participants: Part 1 will recruit women newly operated for breast cancer; Part 2 will recruit women who have completed radiation therapy for breast cancer. Both groups will receive the same intervention and the same information will be captured from all enrolled participants on retention, adherence, and acceptability of the intervention being tested. Outcomes related to the feasibility of the intervention will be collected before and following the 12-week intervention.

Using the PICOT format the trial parameters are:

Population: Women who underwent surgery for breast cancer within the last 8 weeks (part 1) and women who have had surgery and have completed radiation therapy for breast cancer within the past 6 weeks (part 2).

Intervention: Participants will get a leaflet with upper-body rehabilitation exercises and have access to an online rehabilitation platform for the 12-week study period. The platform is a website with videos of upper body rehabilitation exercises, mindfulness sessions and instruction in lymphatic drainage combined with additional information about prevention and early detection of late effects after breast cancer treatment. The intervention will be tailored to each woman with specific upper body exercises based on the baseline arm assessment. The physiotherapist will deliver a leaflet with exercises and educational information to support the engagement in home-based exercises. In addition to this intervention, all participants will be offered the existing rehabilitation program in the trial sites. The programs differ from site to site, but generally include post-surgery upper-body rehabilitation group sessions, general whole body aerobic and resistance training and individual treatment and instruction by a physiotherapist if issues are noted during the group sessions.

Comparison: For this feasibility study, no control group will be used.

Outcome: Outcomes are recruitment rate, adherence and retention, participant satisfaction, capacity/resources and response-rate to the questionnaires concerning intention, attitude, subjective norm, and perceived behavioral control to do home-based exercises, and shoulder function.

Time of intervention: Participants in part 1 will be recruited up to eight weeks after breast cancer surgery, when they start the municipal rehabilitation, and after inclusion followed for 12 weeks. Participants in part 2 will be recruited when the have completed radiation therapy for breast cancer, and after inclusion followed for 12 weeks.

Study conduct:

This study has obtained ethical approval from the Danish National Committee on Health Research Ethics, the Danish Data Protection Agency and has been submitted for ethical approval for the University of British Columbia Clinical Research Ethics Board. The study will be conducted in accordance with the protocol and the Helsinki Declaration. All study participants will sign an informed consent form prior to beginning the study.

Participants:

All patients who have received surgery for breast cancer at the identified clinical sites, and meet the eligibility criteria will be approached to participate in the study. Specifically, women attending the rehabilitation centers in 11 municipalities in Denmark (Copenhagen, Frederiksberg, the 3-municipality collaboration between Gentofte, Rudersdal and Lyngby-Taarbæk, and the 6-municipality collaboration between Herlev, Egedal, Ballerup, Rødovre, Furesø and Gladsaxe) will be recruited. Patients will be eligible and offered to participate if they comply with the inclusion and exclusion criteria.

Outcomes:

Outcomes will be assessed at baseline and end of study. The baseline assessment includes standardized questionnaires and a clinical upper-body assessment. Similar questionnaires will be completed at the 12-week follow up visit.

Primary outcomes: The primary objective of this study is to determine the feasibility and acceptability of this type of online rehabilitation to breast cancer survivors prior to progression to a full RCT. Feasibility will be measured using the four indicators listed below.

Recruitment rate: All reasons for ineligibility or participant refusal to participate will be recorded to explain if any changes should be made to eligibility criteria in future studies.

Retention and Adherence and safety to the intervention: Participants will be asked to record their adherence to their home-based rehabilitation program (i.e. sessions per week) in a logbook on a weekly basis and return the logbook at the end of the study. Program-specific outcomes such as the time spent doing rehabilitation exercises, pain/discomfort during or following the home-based rehabilitation exercises and reasons for discontinuing the rehabilitation program are included in this logbook, as well as participation in other rehabilitation exercise activities, breast cancer-specific group-based rehabilitation sessions or treatment by a physiotherapist. Participant adherence to the home-based exercise prescription will be calculated by the proportion of weeks where the home-based program was performed 5 to 7 times. In addition, the participants' use of the website will be tracked, specifically the website will track the number of times and the duration a participant has been logged onto the website across the 12 weeks. Participants who are enrolled in the study but fail to complete the end of study assessment will be recorded as dropouts. All dropouts will be contacted to determine reasons for non-participation and to collect suggestions for changes. If willing, they will be asked to complete the participant satisfaction questionnaire (see below for details). Feasibility will be defined as a drop out of <10% and adherence of > 75% to the prescribed home-based exercise sessions as determined by reports of performing the home-based program 5 to 7 times weekly in the weekly logbooks.

Participant Satisfaction: At the end of the study data describing participant satisfaction will be collected to answers questions on acceptability. All participants will be given a questionnaire, delivered by Easy Research, and will be asked to rank various aspects of the intervention such as the home-based exercises supported by videos, mode of delivery, software, etc. "as not at all satisfied", "not very satisfied", "somewhat satisfied" or "very satisfied". Feasibility will be defined as >75% of participants reporting they are "very" or "somewhat satisfied" with the intervention.

Capacity/ Resources: The amount of time spent with each participant during the standard upper-body assessments, instruction of the home-based intervention and assistance needed with using the website during the study period will be tracked. We will also record any additional appointments required to teach the home-based rehabilitation program or to assist in using the website.

Secondary outcomes: In addition to the feasibility outcomes, the aim is to examine changes in outcomes of interest that may occur as a result of participation in this 12-week intervention.

Intention, Attitude, Subjective norm, and Perceived behavior control for rehabilitation exercises: To further answers questions on motivation, the participants' reaction to the intervention, intend to use, and perceived appropriateness of the rehabilitation exercises will be answered. Behavioral changes in motivation to do home-based rehabilitation exercises will be measured as this is fundamental to adherence. The study method is theoretically based in the framework of Theory of Planned Behavior and has been validated in measuring motivation for exercise among cancer survivors including breast cancer patients. The Intention, Attitude and Subjective Norm Questionnaire is a 13-item Theory of Planned Behavior questionnaire modified for use with online home-based rehabilitation.

Clinical outcomes in upper-body function: At baseline and after the 12-week intervention, physiotherapists blinded to prior baseline measurements will perform a standard upper-body assessment in all participants. Following measures will be assessed: 1) active shoulder mobility for flexion and external rotation 2) upper body muscle strength using Manual Muscle Testing 3) arm circumference will be measured at five points along the arm using a standardized protocol and measurement tape 4) patient-reported pain and tightness will be measured using a 0-10 VAS scale.

Ability to perform activities of daily living: The self-reported QuickDASH (Disabilities of the Arm, Shoulder, and Hand) is an 11-item questionnaire assessing arm disability affecting multiple arm joints. The QuickDASH will be administered at baseline and at the 12-week follow up visit, and will be used to assess changes in arm function during the study period.

Timeline and proposed sample size:

This study is the first to assess the feasibility of a new online rehabilitation platform. The aim is to start recruitment for the feasibility study from all 11 sites as soon as ethical approval has been obtained. For this feasibility study, the goal is to recruit as many women as possible during an eight-week recruitment period. Following the 12-week intervention, the study is expected to be completed in June 2016.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast cancer
* Part 1 only: Surgery for breast cancer within the past eight weeks (mastectomy or lumpectomy with either sentinel or axillar dissection), including those women with a history of previous surgery for breast cancer, radiation therapy or chemotherapy
* Part 2 only: Completion of surgery and radiation therapy for breast cancer within the past six weeks.
* Home access to internet from stationary computer, lab top or tablet
* Ability to use internet
* Ability to read and understand Danish

Exclusion Criteria:

* Surgery for breast cancer with immediate breast reconstruction
* Diagnosis of primary lymphedema
* Metastatic or inflammatory breast cancer
* Planned use of chemotherapy within the next 6 weeks
* Surgical complications: infection, drainage issues, seroma, hematoma
* Severe physical, cognitive, or psychiatric illness causing inability to follow the study protocol: i.e. severe depression, anxiety, dementia, poor physical health with likely possibility of hospitalization within the next twelve weeks.
* Planned hospitalization or surgery within the next twelve weeks
* Participation in another clinical trial with a rehabilitation or exercise intervention

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2016-02; Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Campbell, PhD, Principal Investigator — University of British Columbia
Locations (6):
- Denmark (6):
  - Tranehaven, Charlottenlund
  - Copenhagen Centre for Cancer and Health, Copenhagen
  - Sundhedscenter Frederiksberg, Frederiksberg
  - Lukas, Hellerup
  - Træningscenteret Møllebo, Lyngby
  - Furesø Kommunes Genoptræningscenter, Værløse

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We had pre-defined recruitment period and not a sample size goal. The recruitment period was 10 weeks for part 1 of the study (recruiting women within 8 weeks of surgery for breast cancer) and 20 weeks for part 2 (recruiting women within 6 weeks of completing radiation therapy for breast cancer).
Groups:
- Part 1: Home-based Rehabilitation: Home-based upper-body rehabilitation with online support
  Participants in both Part 1 and Part 2 received the same home-based upper-body rehabilitation with online support: Participants received written educational material, in which the physiotherapist marked the exercises specifically recommended for the individual patient. In addition, participants were provided with a personal password giving access to the BRECOR website for 12 weeks. The website contains professionally filmed videos of upper-body rehabilitation exercises (joint mobility and muscle strength) and instructions in scar tissue massage and manual lymph drainage. Furthermore, mindfulness sessions and additional information about prevention and early detection of late effects after breast cancer treatment are available on the website.
  On average, participants were asked to complete three rehabilitation exercises a minimum of 4 times weekly with an anticipated duration of approximately 20 minutes.
- Part 2: Home-based Rehabilitation: Participants in both Part 1 and Part 2 received the same home-based upper-body rehabilitation with online support: Participants received written educational material, in which the physiotherapist marked the exercises specifically recommended for the individual patient. In addition, participants were provided with a personal password giving access to the BRECOR website for 12 weeks. The website contains professionally filmed videos of upper-body rehabilitation exercises (joint mobility and muscle strength) and instructions in scar tissue massage and manual lymph drainage. Furthermore, mindfulness sessions and additional information about prevention and early detection of late effects after breast cancer treatment are available on the website.
  On average, participants were asked to complete three rehabilitation exercises a minimum of 4 times weekly with an anticipated duration of approximately 20 minutes.
Period: Overall Study
Arm/Group | Part 1: Home-based Rehabilitation | Part 2: Home-based Rehabilitation
Started | 35 | 24
Completed | 29 | 20
Not Completed | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Part 1: Home-based Rehabilitation; Part 2: Home-based Rehabilitation: Home-based upper-body rehabilitation with online support
  Home-based upper-body rehabilitation with online support: Participants will be given written educational material, in which the physiotherapist marks the exercises specifically recommended for the individual patient. In addition, participants will get a personal password giving access to the BRECOR website for 12 weeks. The website contains professionally filmed videos of upper-body rehabilitation exercises (joint mobility and muscle strength) and instructions in scar tissue massage and manual lymph drainage. Furthermore, mindfulness sessions and additional information about prevention and early detection of late effects after breast cancer treatment are available on the website.
  On average, participants will complete three rehabilitation exercises a minimum of 4 times weekly with an anticipated duration of approximately 20 minutes.
- Total: Total of all reporting groups
Arm/Group | Part 1: Home-based Rehabilitation | Part 2: Home-based Rehabilitation | Total
Number analyzed (Participants) | 35 | 24 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (11.6) | 55.0 (9.9) | 57.8 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 24 | 59
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 35 | 24 | 59
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Rate
Description: This outcome represent the number and proportion (%) of eligible patients who consented to participate in the study. Recruitment was open for 10 weeks for participants in Part 1 and for 20 weeks for participants in Part 2.
Time Frame: 10 weeks for part 1 and 20 weeks for part 2
Population: This was the number of women who were eligible and invited to participate.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Home-based Rehabilitation: Participants in part 1 and part 2 will receive home-based upper-body rehabilitation with online support: Participants will be given written educational material, in which the physiotherapist marks the exercises specifically recommended for the individual patient. In addition, participants will get a personal password giving access to the BRECOR website for 12 weeks. The website contains professionally filmed videos of upper-body rehabilitation exercises (joint mobility and muscle strength) and instructions in scar tissue massage and manual lymph drainage. Furthermore, mindfulness sessions and additional information about prevention and early detection of late effects after breast cancer treatment are available on the website.
  On average, participants will complete three rehabilitation exercises a minimum of 4 times weekly with an anticipated duration of approximately 20 minutes.
Arm/Group | Part 1: Home-based Rehabilitation | Part 2: Home-based Rehabilitation
Number analyzed (Participants) | 44 | 28
Participants | 35 | 24

2. Primary Outcome: Retention
Description: Participants who are enrolled in the study but fail to complete the end of study assessment will be recorded as dropouts. Feasibility will be defined as a drop out of <10%
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Home-based Rehabilitation | Part 2: Home-based Rehabilitation
Number analyzed (Participants) | 35 | 24
Participants | 29 | 20

3. Primary Outcome: Number of Participants Reporting Being "Very Satisfied" or "Somewhat Satisfied" With the Program
Description: At the end of the study data describing participant satisfaction will be collected to answers questions on acceptability. All participants in part 1 and part 2 will be given a questionnaire, delivered by Easy Research, and will be asked to rank various aspects of the intervention such as the home-based exercises supported by videos, mode of delivery, software, etc. "as not at all satisfied", "not very satisfied", "somewhat satisfied" or "very satisfied". Feasibility will be defined as >75% of participants reporting they are "very" or "somewhat satisfied" with the intervention.
Time Frame: 12 weeks
Population: This is the number of participants in part 1 and part 2 who completed the study and who's data was analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Home-based Rehabilitation | Part 2: Home-based Rehabilitation
Number analyzed (Participants) | 29 | 20
Participants | 16 | 12

4. Primary Outcome: Capacity/ Resources
Description: The amount of time spent with each participant during the standard upper-body assessments, instruction of the home-based intervention and assistance needed with using the website during the study period will be tracked. In addition, any additional appointments required to teach the home-based rehabilitation program or to assist in using the website will be recorded. This information will help to determine the resources needed to administer the online component of the home-based program on a larger scale to a broader group of participants. This data was only collected for Part 1.
Time Frame: 12 weeks
Population: The data on capacity was only collected for Part 1 participants and not for part 2.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Part 1: Home-based Rehabilitation | Part 2: Home-based Rehabilitation
Number analyzed (Participants) | 29 | 0
minutes | 92.4 (27.1) |

5. Primary Outcome: Adherence
Description: Participants in part 1 and part 2 were asked to perform the rehabilitation program at least four times weekly for the duration of the study (12 weeks). Adherence was calculated as the number and proportion of participants who reported in a follow-up questionnaire that they had performed four or more weekly sessions. As such, participants who reported to have completed the home-based rehabilitation program 4 times per week were categorized as having adhered to the program. Likewise, participants who reported to have completed the program 3 times or fewer per week were categorized as not having adhered to the program.
Time Frame: 12 weeks
Population: This is the number of participants in part 1 and part 2 who completed the study and who's data was analysed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Home-based Rehabilitation | Part 2: Home-based Rehabilitation
Number analyzed (Participants) | 29 | 20
Participants | 21 | 9

6. Secondary Outcome: Motivation for Rehabilitation Exercises
Description: To answers questions on motivation, the participants' reaction to the intervention, intend to use, and perceived appropriateness of the rehabilitation exercises will be answered. Behavioral changes in motivation to do home-based rehabilitation exercises will be measured as this is fundamental to adherence. The study method is theoretically based in the framework of Theory of Planned Behavior and has been validated in measuring motivation for exercise among cancer survivors including breast cancer patients. The Intention, Attitude and Subjective Norm Questionnaire is a 19-item Theory of Planned Behavior questionnaire modified for use with online home-based rehabilitation. All questions are answered using a 7 point Likert scale and produces effect sizes (Cohen's D). The Theory of Planned Behavior scale is scored on a 0 to 7 scale with a higher score indicating a greater level of motivation.
Time Frame: 12 weeks
Population: In part 1, the subscale "Intention" had too low internal consistency to be included in the analysis. No results are therefore reported for this group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part 1: Home-based Rehabilitation | Part 2: Home-based Rehabilitation
Number analyzed (Participants) | 29 | 20
score on a scale
  Instrumental attitude | 6.45 (0.54) | 6.38 (0.42)
  Affective attitude | 4.82 (1.09) | 4.45 (1.15)
  Intention: number analyzed (Participants) | 0 | 20
  Intention |  | 6.20 (1.12)
  Planning | 5.69 (1.91) | 5.16 (2.00)
  Self-efficacy | 5.90 (1.46) | 5.46 (1.48)
  Perceived behavioral control | 6.09 (1.21) | 5.26 (1.48)
  Subjective norm | 6.34 (0.97) | 5.90 (1.36)

7. Secondary Outcome: Clinical Outcomes in Upper-body Function: Mobility
Description: Active shoulder mobility for flexion and external rotation. Changes from baseline to follow-up (12 weeks later) will be calculated. This data was only collected for participants in part 1.
Time Frame: 12 weeks
Population: A 3-level categorical outcome was applied (not limited, moderately limited, greatly limited).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Home-based Rehabilitation | Part 2: Home-based Rehabilitation
Number analyzed (Participants) | 35 | 0
Participants
  Baseline: Flexion: Not limited | 19 | 0
  Baseline: Flexion: Moderately limited | 13 | 0
  Baseline: Flexion: Greatly limited | 1 | 0
  Baseline: Flexion: Missing | 2 | 0
  End of study: Flexion: number analyzed (Participants) | 29 | 0
  End of study: Flexion: Not limited | 27 | 0
  End of study: Flexion: Moderately limited | 1 | 0
  End of study: Flexion: Greatly limited | 0 | 0
  End of study: Flexion: Missing | 1 | 0
  Baseline: External rotation: Not limited | 17 | 0
  Baseline: External rotation: Moderately limited | 11 | 0
  Baseline: External rotation: Greatly limited | 3 | 0
  Baseline: External rotation: Missing | 4 | 0
  End of study: External rotation: number analyzed (Participants) | 29 | 0
  End of study: External rotation: Not limited | 21 | 0
  End of study: External rotation: Moderately limited | 6 | 0
  End of study: External rotation: Greatly limited | 1 | 0
  End of study: External rotation: Missing | 1 | 0
Statistical Analysis 1: Comparison: Part 1: Home-based Rehabilitation; Test type: Equivalence — Differences (the number of participants in each of the three categories) between baseline and follow-up was calculated using a Wilcoxon signed-rank test. This was a feasibility test and no power calculation was performed; p = 0.05, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Clinical Outcomes in Upper-body Function: Muscle Strength
Description: Upper body muscle strength was tested using Manual Muscle Testing among participants in part 1 only.
Time Frame: 12 weeks
Population: A 3-level categorical outcome was applied (not limited, moderately limited, greatly limited).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Home-based Rehabilitation | Part 2: Home-based Rehabilitation
Number analyzed (Participants) | 35 | 0
Participants
  Baseline: Latissimus Dorsi: Not limited | 25 | 0
  Baseline: Latissimus Dorsi: Moderately limited | 9 | 0
  Baseline: Latissimus Dorsi: Greatly limited | 0 | 0
  Baseline: Latissimus Dorsi: Missing | 1 | 0
  End of study: Latissimus Dorsi: number analyzed (Participants) | 29 | 0
  End of study: Latissimus Dorsi: Not limited | 25 | 0
  End of study: Latissimus Dorsi: Moderately limited | 1 | 0
  End of study: Latissimus Dorsi: Greatly limited | 0 | 0
  End of study: Latissimus Dorsi: Missing | 3 | 0
  Baseline: Serratus Anterior: Not limited | 16 | 0
  Baseline: Serratus Anterior: Moderately limited | 13 | 0
  Baseline: Serratus Anterior: Greatly limited | 1 | 0
  Baseline: Serratus Anterior: Missing | 5 | 0
  End of study: Serratus Anterior: number analyzed (Participants) | 29 | 0
  End of study: Serratus Anterior: Not limited | 16 | 0
  End of study: Serratus Anterior: Moderately limited | 10 | 0
  End of study: Serratus Anterior: Greatly limited | 1 | 0
  End of study: Serratus Anterior: Missing | 2 | 0
  Baseline: Pectoralis Major: Not limited | 13 | 0
  Baseline: Pectoralis Major: Moderately limited | 18 | 0
  Baseline: Pectoralis Major: Greatly limited | 0 | 0
  Baseline: Pectoralis Major: Missing | 4 | 0
  End of study: Pectoralis Major: number analyzed (Participants) | 29 | 0
  End of study: Pectoralis Major: Not limited | 17 | 0
  End of study: Pectoralis Major: Moderately limited | 8 | 0
  End of study: Pectoralis Major: Greatly limited | 0 | 0
  End of study: Pectoralis Major: Missing | 4 | 0
Statistical Analysis 1: Comparison: Part 1: Home-based Rehabilitation; Test type: Equivalence — [test comment as in outcome 7, analysis 1]; p = 0.05, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Clinical Outcomes in Upper-body Function: Arm Circumference
Description: Arm circumference at 5 points along the arm. Changes from baseline will be calculated.
Time Frame: 12 weeks
Population: Handling errors compromised data integrity. Specifically, data was not collected at the end of study time point. This prohibited reporting and analysis of data.
Arm/Group | Part 1: Home-based Rehabilitation | Part 2: Home-based Rehabilitation
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Clinical Outcomes in Upper-body Function: Pain
Description: Patient-reported pain on a 0-10 Visual Analogue Scale in the breast/arm region. A higher score indicates greater level of pain. Changes from baseline will be calculated. This data was only collected for part 1.
Time Frame: 12 weeks
Population: Participants in part 2 did not have a clinical assessment at follow up and this data is therefore not collected for part 2, but only collected for part 1.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Part 1: Home-based Rehabilitation | Part 2: Home-based Rehabilitation
Number analyzed (Participants) | 35 | 0
score on a scale
  Baseline | 1.0 [1.0 to 3.0] |
  Follow up: number analyzed (Participants) | 29 | 0
  Follow up | 1.0 [1.0 to 2.0] |

11. Secondary Outcome: Ability to Perform Activities of Daily Living
Description: QuickDASH (Disabilities of the Arm, Shoulder, and Hand) scores 0 to 100 with higher scores indicating more limitations in upper-body functioning.
Time Frame: 12 weeks
Population: At baseline, 35 participants in part 1 and 20 participants in part 2 completed the QuickDASH questionnaire. At follow-up, 24 participants in part 1 and 17 participants in part 2 completed the questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part 1: Home-based Rehabilitation | Part 2: Home-based Rehabilitation
Number analyzed (Participants) | 35 | 20
score on a scale
  Baseline | 19.8 (13.3) | 13.5 (15.8)
  Follow up: number analyzed (Participants) | 24 | 17
  Follow up | 15.2 (14.8) | 11.0 (8.2)

ADVERSE EVENTS:
Time Frame: The period of time to observe adverse events was 12 weeks from baseline to end of study.
Arm/Group | Part 1: Home-based Rehabilitation | Part 2: Home-based Rehabilitation
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/24
Other Adverse Events (participants affected / at risk) | 0/35 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No